CLINICAL TRIAL: NCT04959006
Title: Investigating the Impact of a Natural Antioxidant Food Product on Exerciseinduced Oxidative Stress in Recreationally Active Participants
Brief Title: Investigating a Natural Antioxidant Food Product on Oxidative Stress in Recreationally Active Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Principal Investigator, Justin Roberts, Associate Professor, Anglia Ruskin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R9039
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Oxidative Stress; Exercise Recovery
Keywords: Antioxidants; Exercise Metabolism; Exercise Nutrition

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to either placebo or antioxidant-rich olive extract in a parallel, double blind manner
Who Masked: Participant, Investigator
Masking Description: Nutritional supplements will be provided in a randomised, double-blinded manner. Both the participants and research testers will be masked from knowing the specifics of the supplement intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Placebo drink - oral bolus (25ml) - colour/taste matched (prune juice/cola/tonic water, 1:1:1 ratio).
  Interventions: Dietary Supplement: Placebo
- Antioxidant supplement (Experimental): Experimental condition -oral bolus (25ml) olive extract drink(https://www.oliphenolia.it/uk/)
  Interventions: Dietary Supplement: Antioxidant supplement

INTERVENTIONS:
Dietary Supplement: Antioxidant supplement — Short term (16d) supplementation of either the antioxidant supplement (Oliphenolia) or placebo. Participants required to consume 2x25ml drinks, one mid-morning, one mid-afternoon between meals.
  Other Names: Oliphenolia
  Arms: Antioxidant supplement
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The aim of this study is to investigate the short term use of olive extract polyphenols on markers of oxidative stress in response to acute endurance exercise in recreationally active, healthy volunteers.The study will be conducted under laboratory conditions following a 16 day supplemental period. Participants will be required to attend the laboratory for a pre-screening/familiarisation trial followed by assessments PRE (baseline, days 1,2) and POST intervention (days 18,19). Across the intervention, participants will maintain habitual dietary intake/ exercise training.

Additionally participants will be randomised in a double-blinded manner to either a placebo or antioxidant-rich supplementation (olive extract water).

It is hypothesised that the polyphenols (antioxidants) found within olive extract drink will enhance markers of recovery to an endurance exercise bout compared with the placebo drink.

DETAILED DESCRIPTION:
There is current scientific interest in the use of fruit and plant-based polyphenol supplementation for exercise recovery. Current inference highlights that acute supplementation (~3d) with >1000mg polyphenols per day may enhance recovery from intensive exercise, with most focus on pomegranate, cocoa, green tea extracts, Montmorency cherry concentrate and blackcurrant food products. However, further research is needed to access impact of natural polyphenols at lower or similar doses for longer time periods (>7d) on endurance based activities and subsequent recovery.

There has also been significant clinical research interest in the properties of waste water produced when cold pressing olives, which has been shown to contain high concentrations of natural polyphenols. Fattoria La Vialla is an Italian-based organic farm producing various products including cold-pressed olive oil. In doing so, they also produce olive extract which is commercially available as 'Oliphenolia'. Whilst several clinical studies have been undertaken using this product, to date there have been no studies investigating the polyphenol potential of olive extract on exercise recovery and subsequent performance.

As such, this study proposes to investigate the short term use of olive extract polyphenols on markers of oxidative stress in response to acute endurance exercise in recreationally active, healthy volunteers. Following a study briefing and provision of written, informed consent, participants will be required to attend the Human Physiology Laboratory at Anglia Ruskin University on 5 occasions as follows:

Session 1 - assessment of metabolic responses to incremental exercise intensity and individual maximal oxygen uptake (VO2max) using a standardised treadmill-based ramp protocol. Measurement of VO2max will be required for assessment of exercise intensity for sessions 2 and 4 (see below). The treadmill protocol to be used is similar to that previously published, involving two graded exercise tests (GXT1 and GXT2). Following a 10min resting period and assessment of baseline measures (e.g. blood pressure, body composition) and a 5min warm up period, GXT1 will involve participants completing ~6 x 4min stages (3mins running, 1 minute passive recovery in which capillary blood sampling for glucose/lactate will be carried out). Starting speeds will be between ~6-10km/h (1 % gradient) with each stage involving speed increments of 1 km/h. Exercise will continue until blood lactate concentration exceeds 4 mMol/L. Following a 10 min rest, GXT 2 will begin at a speed 2 km·h-1 below the previous GXT 1 final speed, with gradient increasing by 1 % each min and continuing until volitional exhaustion. Throughout the test, breath-to-breath analysis (using a Metalyser 3B respiratory analyser) will be undertaken.

Session 2 - Having overnight fasted, and following resting measures (blood pressure, body composition via bioelectrical impedance analysis, 3x4ml blood sample), participants will complete an endurance training session (~75% VO2max for 60mins) on a treadmill. Additional wholeblood samples (3x4ml) will be collected immediately and 1hr post exercise.

Session 3 - Participants will return the next morning (overnight fasted) for a resting blood sample (3x4ml, 24 hours post exercise) and complete the same GXT1 and GXT2 tests carried out in session 1. This will be used to quantify metabolic and recovery indices.

Session 4 and 5 - following a 16 day nutrition product supplementation period, participants will return and complete exercise testing as per sessions 2 and 3.

Nutritional supplementation - all products will be supplied/certified independently via Fattoria La Vialla, Italy. Participants will be randomly assigned in a double-blinded manner to either: i) Experimental condition: 2x25ml olive extract drinks (https://www.oliphenolia.it/uk/) per day for 16 days, taken one mid-morning, one mid-afternoon between meals or ii) matched placebo (2x25ml of prune juice water).

Blood samples - wholeblood samples will be immediately centrifuged with serum allocated into separate cryovials for the analysis of: i) the main polyphenol compound- hydroxytyrosol; ii) a marker of oxidative stress (malondialdehyde, MDA) and iii) key antioxidant enzymes (catalase, superoxide dismutase) and redox status (reduced glutathione (GSH) to oxidized glutathione (GSSG) ratio).

Over the 16 day study period, there will be no dietary restrictions in place (other than following a low polyphenol diet 24 hours prior to each testing session), however participants will need to follow the allocated supplementation and maintain their training program (~3-4 run training sessions per week).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, UK based, above 21 years of age and below 65 years of age
* All participants: No known history (including family history) of heart abnormalities, hypertension, coronary heart disease or diabetes (determined from pre-study health screen questionnaire)
* All participants: Not currently suffering from any musculo-skeletal injury, or any other reason that may prevent participation in cardiovascular exercise
* All participants: Have not suffered from recent viral infections ie: influenza (defined within the prior 2 months)
* All participants (and household members): COVID-19 related - have not suffered with any symptoms associated with Covid-19
* All participants: Not suffering from any known blood related disorders, including blood coagulation abnormalities, or have any adverse reactions to blood taking
* All participants: Not taking any prescribed or over-the-counter medication which may influence exercise training (with the exception of inhalers for exercise induced asthma or contraceptive pill)
* All participants: Not consuming or prepared to refrain from consumption, any commercial supplementation which conflicts with the study parameters ie: antioxidants.
* All participants: no known allergy or intolerance to olives or prune/grape juice.
* Baseline maximal oxygen uptake >25ml/kg/min representative of normal fitness levels (measured during pre-screening)

Exclusion Criteria:

* Anyone below the age of 21 years or above 65 years of age
* All participants: anyone with a known history (including family history) of heart abnormalities, hypertension, coronary heart disease or diabetes (determined from pre-study health screen questionnaire)
* All participants: Anyone suffering from a current musculo-skeletal injury, or any other reason that may prevent participation in cardiovascular exercise
* All participants: those suffering from recent viral infections ie: influenza (defined within the prior 2 months)
* All participants: anyone who has (previously or currently) had any symptoms associated with covid-19 (including household members)
* All participants: Those with known blood related disorders, including blood coagulation abnormalities, or have any adverse reactions to blood taking. This includes any participant who has or potentially has an infectious disease, inc. HIV, and all types of hepatitis.
* All participants: Anyone taking any prescribed or over-the-counter medication which may influence exercise training (with the exception of inhalers for exercise induced asthma or contraceptive pill)
* All participants: Anyone consuming or not prepared to refrain from consumption, any commercial supplementation which conflicts with the study parameters ie: antioxidants
* All participants: anyone with a known allergy or intolerance to olives or prune/grape juice.
* Any not meeting the baseline criteria for maximal oxygen uptake
* FEMALE ONLY: Any participant who is, suspects they may be or becomes pregnant during the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress biomarker | Change from pre (day 1) to post intervention (day 18)
  Blood measure of malondialdehyde, MDA (pmol/ml)
Redox status | Relative change from pre (day 1) to post intervention (day 18)
  Blood measure of reduced glutathione (GSH) to oxidized glutathione (GSSG) (measured in uM)
Endogenous antioxidant enzyme 1 | Relative change from pre (day 1) to post intervention (day 18)
  Blood measure of catalase (mU/ml)
Endogenous antioxidant enzyme 2 | Relative change from pre (day 1) to post intervention (day 18)
  Blood measure of superoxide dismutase (inhibition rate %)
Hydroxytyrosol | Overall change from pre (day 1) to post intervention (day 18)
  Blood measure of hydroxytyrosol (main active ingredient in the antioxidant supplementation, measured in ng/ml)

SECONDARY OUTCOMES:
Submaximal exercise respiratory measures | Relative change from pre (day 1) to post intervention (day 18)
  Assessment of metabolic efficiency via respiratory measures (oxygen, carbon dioxide, both measured in L/min) during steady state exercise
Maximal exercise respiratory measures | Relative change from pre (day 1) to post intervention (day 18)
  Assessment of exercise capacity and tolerance during maximal exercise via respiratory measures (oxygen, carbon dioxide, both measured in L/min)
Body mass | Change from pre (day 1) to post intervention (day 18)
  Assessment of body mass (kg). Body mass and height will be combined to report Body Mass Index (BMI) in kg/m^2
Height | Change from pre (day 1) to post intervention (day 18)
  Assessment of participant height (m). Body mass and height will be combined to report Body Mass Index (BMI) in kg/m^2
Body composition | Change from pre (day 1) to post intervention (day 18)
  Assessment of bodyfat (%) used to derive lean mass (kg) based on total body mass (kg)
Blood pressure | Change from pre (day 1) to post intervention (day 18)
  Assessment of systolic and diastolic blood pressure (measured in mmHg) at rest

CONTACTS AND LOCATIONS:
Overall Officials: Justin Roberts, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- Anglia Ruskin University, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowtell J, Kelly V. Fruit-Derived Polyphenol Supplementation for Athlete Recovery and Performance. Sports Med. 2019 Feb;49(Suppl 1):3-23. doi: 10.1007/s40279-018-0998-x. PMID 30671906
- [Background] Fisher-Wellman K, Bloomer RJ. Acute exercise and oxidative stress: a 30 year history. Dyn Med. 2009 Jan 13;8:1. doi: 10.1186/1476-5918-8-1. PMID 19144121
- [Background] Bloomer RJ, Goldfarb AH, McKenzie MJ. Oxidative stress response to aerobic exercise: comparison of antioxidant supplements. Med Sci Sports Exerc. 2006 Jun;38(6):1098-105. doi: 10.1249/01.mss.0000222839.51144.3e. PMID 16775552
- [Background] James CA, Richardson AJ, Watt PW, Gibson OR, Maxwell NS. Physiological responses to incremental exercise in the heat following internal and external precooling. Scand J Med Sci Sports. 2015 Jun;25 Suppl 1:190-9. doi: 10.1111/sms.12376. PMID 25943670